CLINICAL TRIAL: NCT01621893
Title: Prospective Efficacy Evaluation of Subchondroplasty™ for the Treatment of Defects Associated With Tibial Bone Marrow Lesions
Brief Title: Evaluation of Subchondroplasty™ for Defects Associated With Bone Marrow Lesions
Acronym: SCP
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: KC-SCP-001
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Bone Marrow Edema
Keywords: bone marrow edema; bone marrow defects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- BML of the Knee: Subject has single bone marrow lesion of tibia, single BML of femur, or adjoining BML's of tibia & femur on which a Subchondroplasty procedure is performed
  Interventions: Procedure: Subchondroplasty

INTERVENTIONS:
Procedure: Subchondroplasty
  Other Names: Calcium Phosphate Bone substitute filling of micro fractures

SUMMARY:
Studying long-term changes in a sub-set of patients who undergo the Subchondroplasty procedure including changes in pain, function, and overall health.

DETAILED DESCRIPTION:
This study is designed as a prospective, consecutive series outcomes study. Patients presenting with knee pain associated with bone marrow lesions that meet the inclusion criteria will be eligible to undergo Subchondroplasty procedure. The subjects will be followed for twenty-four (24) months after surgery via office visits and will be contacted once per year for up to 5 years post-operatively and asked questions regarding their pain and functioning to further understand long-term outcomes.. Seventy (70), a ( minimum of sixty-two (62)) patients who meet the inclusion/exclusion criteria will be enrolled in the study. Up to 5 sites will participate in this study. The study is intended to provide an estimate of one-year and two-year clinical success with minimum bias and with sufficient statistical precision to permit meaningful comparison to commonly accepted two-year clinical success rates for currently available treatment alternatives. An improvement of 10 points on the Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscore on the KOOS Scoring System from baseline to 1-year post-operative is considered minimal perceptible clinical improvement and will be used to define the primary clinical success criterion for this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 40-70 of age and skeletally mature
* Subject BMI is < 40
* Subject has experienced pain in knee for at least 3 months
* BML is confirmed on T2 weighted MR Imaging by presence of white signal
* Subject has single BML of tibia, single BML of femur, or adjoining BML's of tibia & femur
* Baseline KOOS pain subscore is ≤65
* Subject's involved knee alignment is defined radiographically as one of the following: Neutral, ≤ to 7 degrees mechanical varus or < 7.5 degrees mechanical valgus
* Subject's ACL and PCL ligaments are intact
* Subject has failed no more than one operative treatment on treatment knee, and none within 6 months prior to enrollment
* Subject is willing and able to sign a written consent form
* The subject has the mental capacity and the willingness to comply with the specified follow-up evaluations, and can be contacted by telephone by the site personnel.

Exclusion Criteria:

* Surgeon deems subject's pain to be primarily related to an alternate condition such as a baker cyst, synovitis, meniscal pathology, or other
* BML caused by acute trauma
* Subject is not neurologically intact (sensory, motor, and reflex deficit)
* Subject is insulin dependent
* Subject has a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for 5 years
* Subject with primary bone tumor in the knee area
* Subject anticipates having a lower extremity surgery other than the investigational surgery during the course of the study
* Subject has a history of substance abuse
* Subject is currently involved in another study or have received investigational product or treatment within the last 30 days
* Subject is pregnant or planning on becoming pregnant during the study period
* Subject is accepting workers' compensation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with single bone marrow edema of the tibia, single bone marrow lesion of the femur or adjoining bone marrow lesions of the tibia and femur (kissing lesions).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Knee Injury Osteoarthritis Outcomes Score (KOOS) Pain Subscore | 1 Year
  Post-operative KOOS pain subsection score at 1-Year follow-up is improved by at least 10 points. The KOOS is a validated instrument which measures knee pain and function using five subscales: pain, symptoms, function in daily living, function in sport and recreation, and quality of life. The instrument consists of 42 standardized questions each having 5 point Likert response scale

SECONDARY OUTCOMES:
Improvement from baseline in KOOS subsection scores | 24 Months
  The KOOS is a validated instrument which measures knee pain and function using five subscales: pain, symptoms, activities of daily living (ADL), function in sport and recreation, and quality of life. The instrument consists of 42 standardized questions each having 5 point Likert response scale.
Improvement in VAS | 24 Months
  The VAS is a validated pain scale. Subjects are asked to rate the amount of pain they have experienced with activity (walking, climbing stairs) for the past week by placing a slash through a 100mm line, which bests describes the pain when 0 is no pain and 100 is worst pain imaginable. Study personnel will measure where the subject placed the mark and transcribe this on an eCRF.
Improvement in Modified Knee Score | 24 Months
  Subjects will be asked to complete the Modified Knee Score pre-operatively and at each follow-up visit. The Modified Knee Score is a validated questionnaire composed of 4 questions to evaluate pain and function primarily before and after knee arthroplasty. The score is based on a maximum 100 points with Excellent = 85-100; Good = 70-84; Fair = 60-69; Poor = <60
Improvement in IKDC | 24 Months
  The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. A score of zero is the lowest level of function or highest level of symptoms to 100, highest level of function and lowest level of symptoms.
Maintenance or improvement in usage (i.e., reduction in usage) of NSAIDs, narcotics, anti-inflammatory medications | 24 Months
  Subjects will be asked pre-operatively what medications are taken as part of their knee treatment and at each follow-up visit, medications taken or currently taking as part of their recovery
Complications or secondary procedures at index site of knee | 24 Months
  Incidence of secondary or revision procedures will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Rothman Institute
Locations (6):
- United States (6):
  - CORE Orthopaedics, Encinitas, California
  - Hinsdale Orthopedics, New Lenox, Illinois
  - Hospital for Joint Disease, New York, New York
  - Rothman Institute, Philadelphia, Pennsylvania
  - Allegheny Orthopaedic Associates, Pittsburgh, Pennsylvania
  - Steadman Hawkins Foundation, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen SB, Hajnik C, Loren GJ, Akhavan S, DeMeo PJ, Wyland DJ, Youm T, Jazrawi LM, Daley RJ, Farr J, Reischling P, Woodell-May JE. Prospective Evaluation of Clinical Outcomes of the Subchondroplasty Procedure for Treatment of Symptomatic Bone Marrow Lesions of the Knee. J Knee Surg. 2025 May;38(6):290-299. doi: 10.1055/a-2501-0910. Epub 2024 Dec 12. PMID 39667406